CLINICAL TRIAL: NCT07212192
Title: Effectiveness of 10% Lidocaine Spray on Relieving Local Pain Caused by Intravenous (IV) Intubation: a Randomized Control Trial
Brief Title: Effectiveness of 10% Lidocaine on Relieving Pain Caused by Intravenous Intubation
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Phenikaa University (Other)
Responsible Party: Principal Investigator, Hoang T.X Huong, Vice - Dean of Nursing Faculty, Phenikaa University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PKA_01
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy
Keywords: Lidocaine; IV pain; C-Section

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 2 (Placebo Comparator): Participants will be given three sprays sterilized saline solution 3 minutes before the interventionist performed the insertion of a catheter into their vein
  Interventions: Combination Product: Sterilized saline solution
- Group 3 (No Intervention): Non intervention will be perform rather than usual care
- Intervention (Experimental): Participants will be given three sprays of 10% Lidocaine (Lidocaine 10% pump spray, Egis) 3 minutes before the interventionist performed the insertion of a catheter into their vein
  Interventions: Drug: Lidocain spray

INTERVENTIONS:
Drug: Lidocain spray — Applying 3 spray of 10% Lidocaine to the IV insertion site in women before their C-section
  Arms: Intervention
Combination Product: Sterilized saline solution — Participants will be given three sprays sterilized saline solution 3 minutes before the interventionist performed the insertion of a catheter into their vein
  Arms: Group 2

SUMMARY:
The goal of this clinical trial is to learn if 10% Lidocaine spray can reduce local pain caused by intravenous (IV) intubation among women. The main questions it aims to answer are:

* Does 10% Lidocaine spray lower the VAS score in participants need intravenous intubation?
* What size effect of 10% Lidocaine spray when patients administered? Researchers will compare 10% Lidocaine spray to a placebo (a look-alike substance that contains no drug) to see if 10% Lidocaine spray works to reduce local pain caused by intravenous (IV) intubation

Participants will:

* Receive 3 spray of 10% Lidocaine at intravenous catheter insertion site before the nurse perform the IV insert procedure
* Assess the pain cause by IV insertion using VAS

DETAILED DESCRIPTION:
Intravenous (IV) cannulation is a technique in which a cannula is placed inside a vein through the patient's skin. It is the most commonly performed procedure in clinical settings. Nevertheless, it is also the second most painful procedure that significantly elevates a patient's anxiety levels. IV is required for every patient before their operation. Managing this pre-operative pain has been listed as an indicator of the quality of anesthesia. As such, various interventions have been conducted to reduce the pain caused by intravenous intubation among patients. Non-pharmacological approaches to reduce this pain include using the flash of light to distract patients, cough tricks, Valsalva manoeuvers, and vapor coolant spray, essential oil . Pharmacological approaches for reducing local pain caused by IV include Lidocaine cream/patch/spray, EMLA (mixture of Lidocaine and Prilocain), diclofenac transdermal, and Piroxicam gel . However, none of these methods exhibited a clear superiority over the others. There is no clear consensus about which method is the best option to relieve pain induced by IV. Among pharmacological approaches, using Lidocaine provides some promising results in reducing pain related to IV insertion. Among the different dosage forms, Lidocaine spray is the most convenient with a fast effect. It is quickly absorption within 1 to 5 minutes. However, inconsistent results have been reported regarding this application . Notably, previous trials conducted in different populations, ages, settings, and needle sizes somewhat cause bias in the results. As such, more trials with rigorous design should be implemented to provide strong evidence to support the role of Lidocaine spray in reducing local paint caused by IV intubation. The objective of this study was to evaluate the effect of Lidocaine spray on relieving local pain caused by intravenous intubation. To ensure a homogeneous population, we chose the participants who were women before their Cesarean section delivery (C-section).

ELIGIBILITY:
Inclusion criteria

* Inclusion criteria comprised participants who were going to undergo a scheduled C-section delivery
* Over 18 years old
* Able to read and write Vietnamese.
* Sign the consent form

Exclusion criteria

• Participants who were emergency cases for going to a C-section delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Pain score | After the nurse insert the IV into the participants
  The Pain score will be measured by a visual analog scale (VAS). This is a validated, subjective measure of pain. It is typically a 10-cm line, used to assess a person's perception of pain, discomfort, or other subjective feelings by having them mark a point on the line that best represents their experience. It ranged from 0 to 10, with 0 meaning "no pain" and 10 meaning "worst pain ever". The greater score, indicate greater pain.

SECONDARY OUTCOMES:
Adverse event | List any side effect of Lidocaine reported by participant or observed by PI within 2 hours after the IV has been inserted
  Side effects cause by Lidocaine

CONTACTS AND LOCATIONS:
Overall Officials: Huong Hoang, PhD, Principal Investigator — Phenikaa University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luangtangvarodom W, Pongrojpaw D, Chanthasenanont A, Pattaraarchachai J, Bhamarapravatana K, Suwannarurk K. The Efficacy of Lidocaine Spray in Pain Relief during Outpatient-Based Endometrial Sampling: A Randomized Placebo-Controlled Trial. Pain Res Treat. 2018 Oct 21;2018:1238627. doi: 10.1155/2018/1238627. eCollection 2018. PMID 30420917
- [Background] Dalvandi A, Ranjbar H, Hatamizadeh M, Rahgoi A, Bernstein C. Comparing the effectiveness of vapocoolant spray and lidocaine/procaine cream in reducing pain of intravenous cannulation: A randomized clinical trial. Am J Emerg Med. 2017 Aug;35(8):1064-1068. doi: 10.1016/j.ajem.2017.02.039. Epub 2017 Feb 27. PMID 28285862
- [Background] Kartufan FF. Padded Dressing with Lidocaine HCL for Reducing Pain during Intravenous Cannulation in Adult Patients: A Randomized Controlled Clinical Trial. Biomed Res Int. 2022 Apr 23;2022:6128557. doi: 10.1155/2022/6128557. eCollection 2022. PMID 35502334
- [Background] Datema J, Veldhuis J, Bekhof J. Lidocaine spray as a local analgesic for intravenous cannulation: a randomized clinical trial. Eur J Emerg Med. 2019 Feb;26(1):24-28. doi: 10.1097/MEJ.0000000000000496. PMID 28799984
- [Background] Basaranoglu G, Basaranoglu M, Erden V, Delatioglu H, Pekel AF, Saitoglu L. The effects of Valsalva manoeuvres on venepuncture pain. Eur J Anaesthesiol. 2006 Jul;23(7):591-3. doi: 10.1017/S0265021506000160. Epub 2006 Mar 1. PMID 16507182
- [Background] Alan N, Khorshid L. Evaluation of Efficacy of Valsalva Maneuver During Peripheral Intravenous Cannulation on Pain. Pain Manag Nurs. 2022 Apr;23(2):220-224. doi: 10.1016/j.pmn.2021.01.013. Epub 2021 Mar 9. PMID 33712356
- [Background] Hocking G, Weightman WM, Smith C, Gibbs NM, Sherrard K. Measuring the quality of anaesthesia from a patient's perspective: development, validation, and implementation of a short questionnaire. Br J Anaesth. 2013 Dec;111(6):979-89. doi: 10.1093/bja/aet284. Epub 2013 Aug 28. PMID 23985532
- [Background] Goudra BG, Galvin E, Singh PM, Lions J. Effect of site selection on pain of intravenous cannula insertion: A prospective randomised study. Indian J Anaesth. 2014 Nov-Dec;58(6):732-5. doi: 10.4103/0019-5049.147166. PMID 25624538
- [Background] Sebbane M, Claret PG, Lefebvre S, Mercier G, Rubenovitch J, Jreige R, Eledjam JJ, de La Coussaye JE. Predicting peripheral venous access difficulty in the emergency department using body mass index and a clinical evaluation of venous accessibility. J Emerg Med. 2013 Feb;44(2):299-305. doi: 10.1016/j.jemermed.2012.07.051. Epub 2012 Sep 13. PMID 22981661

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT07212192/Prot_SAP_000.pdf